CLINICAL TRIAL: NCT03959488
Title: A Phase 2/3 Randomized, Double-blind, Palivizumab-controlled Study to Evaluate the Safety of MEDI8897, a Monoclonal Antibody With an Extended Half-life Against Respiratory Syncytial Virus, in High-risk Children (MEDLEY)
Brief Title: A Study to Evaluate the Safety of MEDI8897 for the Prevention of Medically Attended Respiratory Syncytial Virus(RSV) Lower Respiratory Track Infection (LRTI) in High-risk Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D5290C00005; 2019-000201-69 (EudraCT Number)
Record Dates: First submitted 2019-05-21; First posted 2019-05-22 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory Syncytial Virus Infections; Preterm Infants; Lower Respiratory Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Palivizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MEDI8897 (Experimental): anti-RSV monoclonal antibody with an extended half-life
  Interventions: Drug: MEDI8897
- Palivizumab (Active Comparator): anti-RSV monoclonal antibody
  Interventions: Drug: Palivizumab

INTERVENTIONS:
Drug: MEDI8897 — Anti-RSV monoclonal antibody with an extended half-life
  Arms: MEDI8897
Drug: Palivizumab — Approved anti-RSV monoclonal antibody
  Arms: Palivizumab

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of MEDI8897 compared to palivizumab when administered to preterm infants entering their first RSV season and children with chronic lung disease (CLD) and congenital heart disease (CHD) entering their first and second RSV season.

DETAILED DESCRIPTION:
This study is a pivotal Phase 2/3 randomized, double-blind, palivizumab-controlled study to evaluate the safety, pharmacokinetics (PK), anti-drug antibody (ADA) response, and descriptive efficacy for MEDI8897 in high-risk infants eligible to receive palivizumab when entering their first or second RSV season (Season 1 or Season 2, respectively). Approximately 900 palivizumab-eligible infants entering their first RSV season will be enrolled into one of 2 cohorts: (1) preterm cohort, including approximately 600 preterm infants (≤ 35 weeks gestational age [GA]) without CLD/CHD, or (2) CLD/CHD cohort, including approximately 300 infants with CLD of prematurity or hemodynamically significant CHD. A minimum of 100 infants with hemodynamically significant CHD will be enrolled. Within each cohort, randomization will be stratified by hemisphere (northern, southern) and subject age at the time of Season 1 randomization (≤ 3 months, > 3 to ≤ 6 months, > 6 months).

ELIGIBILITY:
Inclusion criteria

1. For the preterm cohort (excluding subjects with CLD or hemodynamically significant CHD): preterm infants in their first year of life and born ≤ 35 weeks 0 days GA eligible to receive palivizumab in accordance with national or local guidelines, including those with:

   1. Uncomplicated small atrial or ventricular septal defects or patent ductus arteriosus, or
   2. Aortic stenosis, pulmonic stenosis, or coarctation of the aorta alone
2. For the CLD/CHD cohort:

   1. Subjects with CLD - infants in their first year of life and a diagnosis of CLD of prematurity requiring medical intervention/management (ie, supplemental oxygen, bronchodilators, or diuretics) within the 6 months prior to randomization
   2. Subjects with CHD - infants in their first year of life and documented, hemodynamically significant CHD (must be unoperated or partially corrected CHD) Note: Infants with hemodynamically significant acyanotic cardiac lesions must have pulmonary hypertension (≥ 40 mmHg measured pressure in the pulmonary artery) or the need for daily medication to manage CHD
3. Infants who are entering their first RSV season at the time of screening
4. Written informed consent and any locally required authorization (eg, Health Insurance Portability and Accountability Act in the USA, EU Data Privacy Directive in the EU) obtained from the subject's parent(s)/legal representative(s) prior to performing any protocol-related procedures, including screening evaluations
5. Subject's parent(s)/legal representative(s) able to understand and comply with the requirements of the protocol including follow-up and illness visits as judged by the investigator
6. Subject is available to complete the follow-up period, which will be 1 year after Season 1/ Dose 1 for subjects without CLD/CHD, or 1 year after Season 2/Dose 1 (or last replacement dose as applicable for CHD) for subjects with CLD/CHD

Exclusion criteria

1. Any fever (≥ 100.4°F [≥ 38.0°C], regardless of route) or acute illness within 7 days prior to randomization
2. Any history of LRTI or active LRTI prior to, or at the time of, randomization
3. Known history of RSV infection or active RSV infection prior to, or at the time of, randomization
4. Hospitalization at the time of randomization, unless discharge is expected within the 7 days after randomization
5. Requirement for mechanical ventilation, extracorporeal membrane oxygenation, CPAP, or other mechanical respiratory or cardiac support at the time of randomization
6. Anticipated cardiac surgery within 2 weeks after randomization
7. Anticipated survival of < 6 months after randomization
8. Receipt of any investigational drug
9. Known renal impairment
10. Known hepatic dysfunction including known or suspected active or chronic hepatitis infection
11. Clinically significant congenital anomaly of the respiratory tract
12. Chronic seizure, or evolving or unstable neurologic disorder
13. Prior history of a suspected or actual acute life-threatening event
14. Known immunodeficiency, including human immunodeficiency virus (HIV)
15. Mother with HIV infection (unless the child has been proven to be not infected)
16. Any known allergy, including to immunoglobulin products, or history of allergic reaction
17. Receipt of palivizumab or other RSV mAb or any RSV vaccine, including maternal RSV vaccination
18. Receipt of any monoclonal or polyclonal antibody (for example, hepatitis B immune globulin, intravenous immunoglobulin) or anticipated use during the study
19. Any condition that, in the opinion of the investigator, would interfere with evaluation of the study drug or interpretation of subject safety or study results
20. Concurrent enrollment in another interventional study
21. Children of employees of the sponsor, clinical study site, or any other individuals involved with the conduct of the study, or immediate family members of such individuals

Ages: 0 Years to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 925 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2023-01-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (118):
- United States (30):
  - Research Site, Anaheim, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, National City, California
  - Research Site, Paramount, California
  - Research Site, West Covina, California
  - Research Site, Aurora, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, South Bend, Indiana
  - Research Site, West Des Moines, Iowa
  - Research Site, Louisville, Kentucky
  - Research Site, Jackson, Mississippi
  - Research Site, Columbia, Missouri
  - Research Site, Mineola, New York
  - Research Site, Syracuse, New York
  - Research Site, Durham, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Greenville, South Carolina
  - Research Site, Corpus Christi, Texas
  - Research Site, Layton, Utah
  - Research Site, St. George, Utah
  - Research Site, Charlottesville, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Morgantown, West Virginia
- Research Site, Graz, Austria
- Belgium (2):
  - Research Site, Brussels
  - Research Site, Ghent
- Bulgaria (8):
  - Research Site, Montana
  - Research Site, Pazardzhik
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sliven
  - Research Site, Sofia
  - Research Site, Veliko Tarnovo
- Canada (2):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
- Research Site, Prague, Czechia
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- Research Site, Tampere, Finland
- France (9):
  - Research Site, Amiens
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Bron
  - Research Site, Caen
  - Research Site, Créteil
  - Research Site, Grenoble
  - Research Site, Marseille
  - Research Site, Pau
- Germany (3):
  - Research Site, Frankenthal
  - Research Site, Leipzig
  - Research Site, Mannheim
- Hungary (5):
  - Research Site, Baja
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Kecskemét
  - Research Site, Miskolc
- Italy (2):
  - Research Site, Pisa
  - Research Site, Verona
- Japan (6):
  - Research Site, Fukui-shi
  - Research Site, Fukuoka
  - Research Site, Kitakyusyu-shi
  - Research Site, Maebashi
  - Research Site, Saitama Shi
  - Research Site, Setagaya-ku
- Latvia (2):
  - Research Site, Jēkabpils
  - Research Site, Riga
- Research Site, Kaunas, Lithuania
- Mexico (2):
  - Research Site, Cuernavaca
  - Research Site, México
- Research Site, Christchurch, New Zealand
- Poland (4):
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Wroclaw
- Russia (5):
  - Research Site, Kazan'
  - Research Site, Novosibirsk
  - Research Site, Perm
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- South Africa (4):
  - Research Site, Cape Town
  - Research Site, Johannesburg
  - Research Site, Pretoria
  - Research Site, Soweto
- South Korea (3):
  - Research Site, Ansan-si
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (10):
  - Research Site, Alicante
  - Research Site, Boadilla del Monte
  - Research Site, Elche
  - Research Site, Leganés
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Pozuelo de Alarcón
  - Research Site, Sant Cugat del Vallès
  - Research Site, Tarragona
- Research Site, Stockholm, Sweden
- Turkey (Türkiye) (3):
  - Research Site, Adana
  - Research Site, Izmir
  - Research Site, Kocaeli
- Ukraine (7):
  - Research Site, Chernivtsі
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv Region
  - Research Site, Odesa
  - Research Site, Sumy
  - Research Site, Vinnytsia
- United Kingdom (3):
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Domachowske J, Madhi SA, Simoes EAF, Atanasova V, Cabanas F, Furuno K, Garcia-Garcia ML, Grantina I, Nguyen KA, Brooks D, Chang Y, Leach A, Takas T, Yuan Y, Griffin MP, Mankad VS, Villafana T; MEDLEY Study Group. Safety of Nirsevimab for RSV in Infants with Heart or Lung Disease or Prematurity. N Engl J Med. 2022 Mar 3;386(9):892-894. doi: 10.1056/NEJMc2112186. No abstract available. PMID 35235733
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5290C00005&attachmentIdentifier=7817621f-6d8e-41e6-a839-c1ccdfed21c7&fileName=d5290c00005-study-synopsis.pdf&versionIdentifier=
- See also: MEDLEY Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5290C00005&attachmentIdentifier=ba02bb70-712d-4844-908a-a17816e1e918&fileName=D5290C00005-Protocol.pdf&versionIdentifier=
- See also: Statistical Analysis Plan (SAP) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5290C00005&attachmentIdentifier=1ed84f06-335c-4887-8739-15ccaa840cb3&fileName=D5290C00005-SAP.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In the overall population, 925 infants (615 in preterm cohort, 310 in CLD/CHD cohort) were enrolled from 25 countries and randomized (2:1) to MEDI8897 (n = 616) or palivizumab (n = 309). Of the 310 subjects in the Season 1 CLD/CHD cohort, 262 continued into the Season 2 phase of the study.
Groups:
- MEDI8897: Subjects who were randomized to MEDI8897 group in Season 1
- Palivizumab: Subjects who were randomized to Palivizumab group in Season 1
- MEDI8897/MEDI8897: CHD/CLD subjects who were randomized to MEDI8897 group in Season 1 and remained in MEDI8897 group in Season 2.
- Palivizumab/MEDI8897: CHD/CLD subjects who were randomized to Palivizumab group in Season 1 and re-randomized to MEDI8897 group in Season 2
- Palivizumab/Palivizumab: CLD/CHD subjects who were randomized to Palivizumab group in Season 1 and re-randomized to Palivizumab group in Season 2
Period: Season 1
Arm/Group | MEDI8897 | Palivizumab | MEDI8897/MEDI8897 | Palivizumab/MEDI8897 | Palivizumab/Palivizumab
Started | 616 | 309 | 0 | 0 | 0
Completed | 543 | 263 | 0 | 0 | 0
Not Completed | 73 | 46 | 0 | 0 | 0
Not completed — Other | 6 | 7 | 0 | 0 | 0
Not completed — Withdrawal by parent/guardian | 43 | 28 | 0 | 0 | 0
Not completed — Due to COVID-19 pandemic | 2 | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 17 | 7 | 0 | 0 | 0
Not completed — Death | 5 | 1 | 0 | 0 | 0
Period: Season 2
Arm/Group | MEDI8897 | Palivizumab | MEDI8897/MEDI8897 | Palivizumab/MEDI8897 | Palivizumab/Palivizumab
Started (Only CHD/CLD subjects who completed Season 1 continued into Season 2 phase of the study) | 0 | 0 | 180 | 40 | 42
Completed | 0 | 0 | 174 | 39 | 40
Not Completed | 0 | 0 | 6 | 1 | 2
Not completed — Other | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by parent/guardian | 0 | 0 | 3 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MEDI8897 | Palivizumab | MEDI8897/MEDI8897 | Palivizumab/MEDI8897 | Palivizumab/Palivizumab | Total
Number analyzed (Participants) | 616 | 309 | 180 | 40 | 42 | 1187
Age, Continuous [Mean (Standard Deviation); unit: Months] — Age at Season 1 randomization for Season 1 participants Population: This summary is for Season 1 participants only
  Months
    Age at randomization (months): number analyzed (Participants) | 616 | 309 | 0 | 0 | 0 | 925
    Age at randomization (months) | 3.947 (2.5513) | 3.840 (2.4608) |  |  |  | 3.911 (2.5206)
Age, Continuous [Mean (Standard Deviation); unit: Months] — Age at first dose of Season 2 for Season 2 participants Population: This summary is for Season 2 participants only
  Months
    Age at first dose of Season 2 (Months): number analyzed (Participants) | 0 | 0 | 180 | 40 | 42 | 262
    Age at first dose of Season 2 (Months) |  |  | 16.772 (2.7141) | 16.598 (2.4335) | 16.132 (2.1040) | 16.643 (2.5857)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex summary for Season 1 participants Population: Sex summary for Season 1 participants
  Participants
    number analyzed (Participants) | 616 | 309 | 0 | 0 | 0 | 925
    Female | 297 | 133 | 0 | 0 | 0 | 430
    Male | 319 | 176 | 0 | 0 | 0 | 495
Sex: Female, Male [Count of Participants; unit: Participants] — Sex summary for Season 2 participants Population: Sex summary for Season 2 participants only
  Participants
    number analyzed (Participants) | 0 | 0 | 180 | 40 | 42 | 262
    Female | 0 | 0 | 81 | 15 | 15 | 111
    Male | 0 | 0 | 99 | 25 | 27 | 151
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race summary for Season 1 participants Population: Race summary for Season 1 participants only
  Participants
    number analyzed (Participants) | 616 | 309 | 0 | 0 | 0 | 925
    American Indian or Alaska Native | 11 | 5 | 0 | 0 | 0 | 16
    Asian | 36 | 14 | 0 | 0 | 0 | 50
    Native Hawaiian or Other Pacific Islander | 4 | 1 | 0 | 0 | 0 | 5
    Black or African American | 59 | 29 | 0 | 0 | 0 | 88
    White | 483 | 249 | 0 | 0 | 0 | 732
    More than one race | 6 | 4 | 0 | 0 | 0 | 10
    Unknown or Not Reported | 17 | 7 | 0 | 0 | 0 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race summary for Season 2 participants Population: Race summary for Season 2 participants only
  Participants
    number analyzed (Participants) | 0 | 0 | 180 | 40 | 42 | 262
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 10 | 3 | 2 | 15
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 1
    Black or African American | 0 | 0 | 9 | 2 | 1 | 12
    White | 0 | 0 | 152 | 35 | 38 | 225
    More than one race | 0 | 0 | 3 | 0 | 1 | 4
    Unknown or Not Reported | 0 | 0 | 5 | 0 | 0 | 5
Congenital heart disease [Count of Participants; unit: Participants] — CHD summary for Season 1 participants Population: CHD summary for Season 1 participants only
  Participants
    number analyzed (Participants) | 616 | 309 | 0 | 0 | 0 | 925
    Yes | 70 | 34 | 0 | 0 | 0 | 104
    No | 546 | 275 | 0 | 0 | 0 | 821
Congenital heart disease [Count of Participants; unit: Participants] — CHD summary for Season 2 participants Population: CHD summary for Season 2 participants only
  Participants
    number analyzed (Participants) | 0 | 0 | 180 | 40 | 42 | 262
    Yes | 0 | 0 | 56 | 14 | 11 | 81
    No | 0 | 0 | 124 | 26 | 31 | 181
Chronic lung disease [Count of Participants; unit: Participants] — CLD summary for Season 1 participants Population: CLD summary for Season 1 participants only
  Participants
    number analyzed (Participants) | 616 | 309 | 0 | 0 | 0 | 925
    Yes | 147 | 70 | 0 | 0 | 0 | 217
    No | 469 | 239 | 0 | 0 | 0 | 708
Chronic lung disease [Count of Participants; unit: Participants] — CLD summary for Season 2 participants Population: CLD summary for Season 2 participants only
  Participants
    number analyzed (Participants) | 0 | 0 | 180 | 40 | 42 | 262
    Yes | 0 | 0 | 132 | 25 | 32 | 189
    No | 0 | 0 | 48 | 15 | 10 | 73

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of MEDI8897 as Assessed by the Occurrence of All Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) and Adverse Events of Special Interest (AESIs) and New Onset Chronic Disease (NOCD)
Description: Safety and tolerability of MEDI8897 will be assessed by the occurrence of all treatment-emergent adverse events (TEAEs), treatment-emergent serious adverse events (TESAEs) , adverse events of special interest (AESIs), and new onset chronic diseases (NOCDs)
Time Frame: 360 days post first dose
Population: As-treated population
Measure: Count of Participants; unit: Participants
Groups:
- MEDI8897: Subjects who received MEDI8897 in Season 1
- Palivizumab: Subjects who received Palivizumab in Season 1
- Palivizumab/Palivizumab: CHD/CLD subjects who were randomized to Palivizumab group in Season 1 and re-randomized to Palivizumab group in Season 2.
Arm/Group | MEDI8897 | Palivizumab | MEDI8897/MEDI8897 | Palivizumab/MEDI8897 | Palivizumab/Palivizumab
Number analyzed (Participants) | 614 | 304 | 180 | 40 | 42
Participants
  TEAE | 444 | 215 | 130 | 31 | 29
  TESAE | 80 | 38 | 23 | 4 | 2
  AESI | 3 | 0 | 1 | 0 | 0
  NOCD | 3 | 0 | 1 | 0 | 0

2. Secondary Outcome: Serum Concentrations of MEDI8897 and Palivizumab
Description: Summary of individual MEDI8897 and palivizumab serum concentration data by treatment group along with descriptive statistics.
Time Frame: Day 15, Day 31, Day 151 post first dose in Season 1 and Season 2
Population: As-treated population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Groups:
- Palivizumab/MEDI8897: CLD/CHD subjects who were randomized to Palivizumab group in Season 1 and re-randomized to MEDI8897 group in Season 2
Arm/Group | MEDI8897 | Palivizumab | MEDI8897/MEDI8897 | Palivizumab/MEDI8897 | Palivizumab/Palivizumab
Number analyzed (Participants) | 614 | 304 | 180 | 40 | 42
ug/mL
  Serum concentrations of MEDI8897 and Palivizumab at Day 15: number analyzed (Participants) | 306 | 167 | 78 | 20 | 23
  Serum concentrations of MEDI8897 and Palivizumab at Day 15 | 104.75 (61.8) | 66.43 (55.7) | 149.38 (169.2) | 97.70 (302.0) | 59.62 (102.4)
  Serum concentrations of MEDI8897 and Palivizumab at Day 31: number analyzed (Participants) | 262 | 119 | 90 | 18 | 16
  Serum concentrations of MEDI8897 and Palivizumab at Day 31 | 85.35 (74.2) | 48.10 (50.0) | 89.71 (369.5) | 124.89 (256.1) | 57.77 (56.3)
  Serum concentrations of MEDI8897 and Palivizumab at Day 151: number analyzed (Participants) | 467 | 238 | 164 | 38 | 38
  Serum concentrations of MEDI8897 and Palivizumab at Day 151 | 25.38 (58.8) | 101.56 (65.6) | 39.86 (145.9) | 37.95 (118.6) | 67.66 (111.4)

3. Secondary Outcome: Incidence of Anti-drug Antibody (ADA) to MEDI8897 and Palivizumab in Serum
Description: Incidence of ADA to MEDI8897 and palivizumab as assessed by the percentage of participants with any post-baseline ADA positive by treatment group.
Time Frame: 360 days post first dose
Population: Participants in as-treated population and with at least 1 post-baseline ADA sample
Measure: Number; unit: Percentage of participants
Groups:
- MEDI8897/MEDI8897: CHD/CLD subjects who were randomized to MEDI8897 group in Season 1 and remained in MEDI8897 group in Season 2. Cumulative ADA data of Season 1 + Season 2 is reported.
- Palivizumab/Palivizumab: CHD/CLD subjects who were randomized to Palivizumab group in Season 1 and re-randomized to Palivizumab group in Season 2. Cumulative ADA data of Season 1 + Season 2 is reported.
Arm/Group | MEDI8897 | Palivizumab | MEDI8897/MEDI8897 | Palivizumab/MEDI8897 | Palivizumab/Palivizumab
Number analyzed (Participants) | 587 | 289 | 180 | 40 | 42
Percentage of participants | 5.8 | 6.9 | 11.7 | 2.5 | 14.3

4. Secondary Outcome: Incidence of Medically Attended Lower Respiratory Track Infection (LRTI) and Hospitalization Due to Reverse Transcriptase Chain Reaction (RT-PCR) Confirmed Respiratory Syncytial Virus (RSV) Through 150 Days Post First Dose
Description: Incidence of medically attended LRTI (inpatient and outpatient) due to RT-PCR-confirmed RSV through 150 days after Dose 1 for season 1 and season 2. Incidence of LRTI hospitalizations due to RT-PCR-confirmed RSV through 150 days after Dose 1 for season 1 and season 2.
Time Frame: 150 days post first dose
Population: ITT population
Measure: Number; unit: Percentage of participants
Arm/Group | MEDI8897 | Palivizumab | MEDI8897/MEDI8897 | Palivizumab/MEDI8897 | Palivizumab/Palivizumab
Number analyzed (Participants) | 616 | 309 | 180 | 40 | 42
Percentage of participants
  Incidence of medically attended RSV LRTI through 150 days post first dose, % | 0.6 | 1.0 | 0 | 0 | 0
  Incidence of medically attended RSV LRTI with hospitalization through 150 days post first dose, % | 0.3 | 0.6 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Through 360 days post first dose of Season 1 for MEDI8897 and Palivizumab groups, through 360 days post first dose of Season 2 for MEDI8897/MEDI8897, MEDI8897/Palivizumab, and Palivizumab/Palivizumab groups.
Description: TEAEs of Season 1 are reported for MEDI8897 and Palivizumab groups. TEAEs of Season 2 are reported for MEDI8897/MEDI8897, MEDI8897/Palivizumab, and Palivizumab/Palivizumab groups.
  Adverse events are reported based on as-treated population. Participants who were randomized and not dosed are not included in adverse event summaries.
Groups:
- MEDI8897/MEDI8897: CHD/CLD subjects who received MEDI8897 in both Season 1 and Season 2.
- Palivizumab/MEDI8897: CLD/CHD subjects who received palivizumab in Season 1 and MEDI8897 in Season 2.
- Palivizumab/Palivizumab: CLD/CHD subjects who received Palivizumab in both Season 1 and Season 2.
Arm/Group | MEDI8897 | Palivizumab | MEDI8897/MEDI8897 | Palivizumab/MEDI8897 | Palivizumab/Palivizumab
All-Cause Mortality (participants affected / at risk) | 5/614 | 1/304 | 0/180 | 0/40 | 0/42
Serious Adverse Events (participants affected / at risk) | 80/614 | 38/304 | 23/180 | 4/40 | 2/42
Other Adverse Events (participants affected / at risk) | 435/614 | 211/304 | 129/180 | 31/40 | 29/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI8897 (N=614) | Palivizumab (N=304) | MEDI8897/MEDI8897 (N=180) | Palivizumab/MEDI8897 (N=40) | Palivizumab/Palivizumab (N=42)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Crying (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 11 (11) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dacryocystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 6 (6) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Lower respiratory tract infection viral (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningitis aseptic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metapneumovirus bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rotavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scrotal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheterisation cardiac (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeding disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeding intolerance (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Underweight (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotonia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemic hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Craniosynostosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diaphragm muscle weakness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infantile apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pulmonary artery stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertensive crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fallot's tetralogy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Social problem (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Social stay hospitalisation (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cyanosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular septal defect (Congenital, familial and genetic disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinopathy of prematurity (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI8897 (N=614) | Palivizumab (N=304) | MEDI8897/MEDI8897 (N=180) | Palivizumab/MEDI8897 (N=40) | Palivizumab/Palivizumab (N=42)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 29 (33) | 11 (12) | 10 (12) | 2 (3) | 7 (7)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysbiosis (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyschezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 3 (4) | 2 (3) | 3 (5) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces pale (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 1 (1)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 13 (13) | 9 (9) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infantile colic (Gastrointestinal disorders) | 9 (9) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Infantile spitting up (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Teething (Gastrointestinal disorders) | 31 (35) | 16 (19) | 7 (7) | 0 (0) | 2 (2)
Tongue erythema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 15 (17) | 11 (14) | 6 (7) | 4 (5) | 3 (8)
Calcinosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Developmental delay (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug tolerance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug withdrawal syndrome (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever neonatal (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incarcerated hernia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Medical device site irritation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site rash (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 81 (109) | 43 (57) | 23 (37) | 9 (12) | 6 (14)
Secretion discharge (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaccination site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaccination site reaction (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaccination site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site urticaria (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sphincter of oddi dysfunction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 6 (6) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Milk allergy (Immune system disorders) | 6 (6) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Nutritional supplement allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenoiditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Adenovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anal fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial blepharitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 22 (27) | 9 (12) | 9 (11) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 20 (28) | 10 (16) | 7 (7) | 4 (7) | 1 (1)
Covid-19 (Infections and infestations) | 8 (8) | 2 (2) | 14 (14) | 3 (3) | 5 (5)
Candida infection (Infections and infestations) | 2 (2) | 3 (5) | 1 (1) | 0 (0) | 0 (0)
Candida nappy rash (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 25 (31) | 10 (12) | 11 (11) | 1 (1) | 3 (3)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Coronavirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Croup infectious (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dacryocystitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis infected (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 12 (12) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 5 (8) | 5 (6) | 2 (3) | 1 (1) | 2 (2)
Enterobiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Enterovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Exanthema subitum (Infections and infestations) | 9 (9) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 7 (7) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 19 (21) | 15 (15) | 11 (19) | 1 (1) | 2 (3)
Gastroenteritis adenovirus (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis sapovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 2 (2) | 4 (4) | 2 (2) | 0 (0)
Gastroenteritis yersinia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal bacterial overgrowth (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital infection fungal (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Giardiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 15 (15) | 6 (6) | 9 (9) | 0 (0) | 2 (2)
Herpes virus infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Human herpesvirus 6 infection (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 11 (12) | 7 (12) | 3 (4) | 2 (2) | 1 (1)
Laryngopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lice infestation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac septal hypertrophy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 18 (21) | 10 (13) | 1 (3) | 3 (4) | 0 (0)
Lower respiratory tract infection viral (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 57 (84) | 39 (50) | 26 (55) | 7 (16) | 9 (15)
Oral candidiasis (Infections and infestations) | 10 (10) | 6 (7) | 3 (3) | 0 (0) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 27 (37) | 11 (14) | 12 (16) | 3 (3) | 2 (3)
Otitis media acute (Infections and infestations) | 16 (20) | 14 (18) | 11 (19) | 5 (6) | 2 (4)
Otitis media chronic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Otitis media viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otosalpingitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Parasitic gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 23 (29) | 8 (8) | 7 (9) | 2 (2) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Low cardiac output syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia parainfluenzae viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pustule (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyoderma (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 75 (109) | 40 (64) | 29 (38) | 6 (8) | 6 (16)
Roseola (Infections and infestations) | 8 (8) | 5 (5) | 3 (3) | 1 (1) | 2 (2)
Rotavirus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Salmonellosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Skin candida (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subglottic laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superinfection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suspected covid-19 (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Right atrial dilatation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 3 (3) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 148 (235) | 77 (131) | 48 (86) | 8 (12) | 9 (26)
Urinary tract infection (Infections and infestations) | 6 (8) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 5 (5) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Viral pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Viral rash (Infections and infestations) | 7 (7) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Viral rhinitis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 33 (42) | 14 (15) | 14 (18) | 8 (8) | 2 (2)
Vulvitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Yersinia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accidental exposure to product (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chillblains (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia neonatal (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foreign body in respiratory tract (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Penis injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radial head dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Re-opening of ductus arteriosus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tongue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth avulsion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 25 (36) | 19 (25) | 1 (1) | 0 (0) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood albumin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body temperature abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anomalous pulmonary venous connection (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronavirus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crystal urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Echocardiogram (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterovirus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemophilus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head circumference abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Human rhinovirus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sars-cov-2 test negative (Investigations) | 19 (40) | 10 (15) | 4 (10) | 3 (5) | 1 (1)
Sars-cov-2 test positive (Investigations) | 4 (4) | 3 (3) | 4 (4) | 1 (1) | 2 (2)
Weight abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Feeding disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeding intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brachycephaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Underweight (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight gain poor (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Zinc deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebellar hypoplasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Growth failure (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myosclerosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rickets (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral ventricle dilatation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral palsy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diplegia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dystonia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotonia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infant irritability (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cleft palate (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Motor developmental delay (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Posthaemorrhagic hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Speech disorder developmental (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Congenital choroid plexus cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug dependence (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 6 (11) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep terror (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staring (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Congenital nystagmus (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vesicoureteric reflux (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enlarged clitoris (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital labial adhesions (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scrotal dermatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Congenital oral malformation (Congenital, familial and genetic disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 6 (7) | 6 (6) | 0 (0) | 0 (0)
Cough variant asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cryptorchism (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 41 (53) | 13 (16) | 4 (5) | 1 (1) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (5) | 0 (0) | 0 (0) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertensive crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystic fibrosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 23 (28) | 12 (14) | 14 (25) | 4 (6) | 2 (4)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne infantile (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asteatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Butterfly rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 7 (8) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmorphism (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 14 (15) | 7 (7) | 3 (4) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 11 (12) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 28 (29) | 6 (6) | 8 (9) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 14 (15) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 14 (14) | 11 (14) | 4 (4) | 0 (0) | 1 (1)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema infantile (Skin and subcutaneous tissue disorders) | 10 (11) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid ptosis congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema toxicum neonatorum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 18 (18) | 11 (12) | 1 (1) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 21 (21) | 9 (9) | 4 (4) | 2 (2) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Rash neonatal (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Urticaria papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 5 (5) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenoidectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dacryocystorhinostomy (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear tube insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrostomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myringotomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orchidopexy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tongue tie operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Capillary fragility (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cyanosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngomalacia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricle outflow tract obstruction (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Plagiocephaly (Congenital, familial and genetic disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Vascular malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neurosensory hypoacusis (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Noninfective myringitis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anisocoria (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anisometropia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Astigmatism (Eye disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Choroidal effusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye allergy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye discharge (Eye disorders) | 1 (2) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Eye inflammation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Monocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid function disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heterophoria (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypermetropia (Eye disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammation of lacrimal passage (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital swelling (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinopathy of prematurity (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Strabismus (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal erythema (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal fissure haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankyloglossia acquired (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 37 (39) | 20 (28) | 5 (5) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/88/NCT03959488/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/88/NCT03959488/SAP_001.pdf